CLINICAL TRIAL: NCT04162327
Title: A Phase Ia/Ib, Open-label, Multicenter, Dose-escalation Study Evaluating the Safety, Tolerability, and Potential Efficacy of IBI315, an Anti-HER2/PD-1 Bi-specific Antibody in Patients With HER2-expressing Advanced Solid Tumor
Brief Title: A Phase Ia/Ib Study of IBI315 in Patients With HER2-expressing Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI315A101
Record Dates: First submitted 2019-10-31; First posted 2019-11-14 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ia stage - IBI315 Dose escalation (Experimental)
  Interventions: Drug: IBI315
- Ib stage - IBI315 monotherapy (Experimental)
  Interventions: Drug: IBI315

INTERVENTIONS:
Drug: IBI315 — Patients will receive IBI315 until disease progression, intolerability, informed consent withdraw, or other reasons leading to treatment discontinue.
  Arms: Ia stage - IBI315 Dose escalation
Drug: IBI315 — Patients will receive IBI315 RP2D until disease progression,intolerability, informed consent withdraw, or otherreasons leading to treatment discontinue.
  Arms: Ib stage - IBI315 monotherapy

SUMMARY:
The primary objective of this phase I study is to evaluate the safety and potential efficacy and to determine the recommended phase 2 dose (RP2D) of IBI315, a HER2/PD-1 bi-specific antibody in patients with advanced solid tumors

DETAILED DESCRIPTION:
This phase Ia/Ib, open-label, multicenter study has two stages. The Ia stage is a dose-escalation study that will focus on safety, tolerability, efficacy and RP2D . Patients with HER2-expressing advanced solid tumor who failed from previous standard of care will be enrolled in the phase Ia study. DLT observation period is 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Written (signed) informed consent.
* Life expectancy ≥12 weeks.
* Patients with HER2-expressing advanced solid tumor who failed on current standard of care
* According to RECIST 1.1, at least one measurable lesion (radiation-naïve) exists.
* ECOG performance status 0-1.
* Adequate organ and marrow function evaluated by laboratory tests as follow:

  * CBC: absolute neutrophil count (ANC) ≥ 1.0×109/L (Ia stage) or 1.5×109/L (Ib stage); Platelet (PLT) ≥ 75×109/L; Hemoglobin (HGB) ≥ 9.0g/L;
  * Liver function: Total bilirubin (TBIL) ≤ 1.5×upper limit of normal value (ULN) for patients without hepatic metastases, ≤ 2×ULN for patients with hepatic metastases or Gilbert syndrome; Alanine aminotransferase (ALT) ≤ 2.5×ULN; Aspartate transferase (AST) ≤ 2.5×ULN;
  * Renal function: Clearance of creatinine (CCr) by Cockcroft-Gault formula or 24-hour urine collection ≥ 50ml/min;
  * Urinalysis: urine protein < 2+ or urine protein in 24-hour urine collection < 1g;
  * Coagulation function: activated partial thromboplastin time (APTT）≤ 1.5×ULN; international normalized ratio (INR）≤ 1.5
* left ventricular ejection fraction (LVEF) ≥ 50% by echocardiography;
* Accumulative exposure to doxorubicin ≤ 360mg/m2; accumulative exposure to epirubicin ≤ 720mg/m2;
* Agree to use an approved contraceptive method during the treatment period, until 180 days after last dose of treatment.
* Post-menopause female subject or pre-menopause female with negative HCG level in urine or blood.

Exclusion Criteria:

* Any greater than NCI CTCAE 0/1 adverse event exists within 4 weeks before enrollment, not including hair loss and fatigue;
* Received major surgery or having unhealed wound, ulcer, or bone fracture;• Received whole pelvic radiation;
* Plan to receive any other anti-cancer therapy not specified in the protocol, except for palliative radiotherapy;
* CNS metastasis, spinal compression, or carcinomatous meningitis
* Active autoimmune disease or inflammatory disorders.
* Primary immunodeficiency diseases;
* Pregnant or breast-feeding female.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | up to 9 months
Maximum plasma concentration (Cmax) | up to 9 months
Terminal elimination half-life (T1/2) | up to 9 months
Apparent volume of distribution (Vd) | up to 9 months

SECONDARY OUTCOMES:
Evaluate receptor occupancy (RO) following single-dose or multi-dose of IBI315 | up to 9 months
The percentage of participants with anti-drug antibody (ADA) positive after dosing IBI315 | up to 9 months
The percentage of participants with neutralizing antibody (NAb) positive after dosing IBI315 | up to 9 months

OTHER OUTCOMES:
Evaluate the efficacy in participants with different expression level of HER2 in tumor tissue | up to 9 months
Evaluate the efficacy in participants with different expression level of PD-L1 in tumor tissue | up to 9 months
Evaluate the efficacy in participants with different expression level of tumor infiltrating lymphocyte (TILs) | up to 9 months
Evaluate the efficacy in participants with different subtype of immune cells in peripheral blood | up to 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- The 307th Hospital of Chinese People's Liberation Army, Beijing, China